CLINICAL TRIAL: NCT06386991
Title: Evaluation of the Effects of Different Irrigation Solutions Used in Regenerative Endodontic Treatment of Lower Molars With Open Necrotic Apexes on Postoperative Pain and Lesion Healing
Brief Title: Effect of Different Irrigation Solutions on Postoperative Pain and Lesion Healing
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ipek Eraslan Akyuz, research assistant, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/206
Record Dates: First submitted 2024-04-11; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Endodontic Disease
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Edetic Acid; Citric Acid; Etidronic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ethylenediamine tetraacetic acid (EDTA) (Active Comparator): Regenerative endodontic treatments require the use of irrigation solutions to break down inorganic and organic tissue residues in the root canals. Sodium hypochlorite (NaOCl) and Ethylenediamine tetraacetic acid (EDTA)will be used when disinfecting root canals. (GROUP 1)
  Interventions: Other: Using ethylenediaminetetraacetic acid (EDTA), citric acid ((MONO/ANH) and etidronic acid (HEBP) to clean root canals during regenerative endodontic treatments
- CITRIC ACID (MONO/ANH) (Active Comparator): Regenerative endodontic treatments require the use of irrigation solutions to break down inorganic and organic tissue residues in the root canals. Sodium hypochlorite (NaOCl) and CITRIC ACID (MONO/ANH) be used when disinfecting root canals. (GROUP 2)
  Interventions: Other: Using ethylenediaminetetraacetic acid (EDTA), citric acid ((MONO/ANH) and etidronic acid (HEBP) to clean root canals during regenerative endodontic treatments
- ETİDRONİC ACID (HEBP) (Active Comparator): Regenerative endodontic treatments require the use of irrigation solutions to break down inorganic and organic tissue residues in the root canals. Sodium hypochlorite (NaOCl) and ETİDRONİC ACID (HEBP) be used when disinfecting root canals. (GROUP 3)
  Interventions: Other: Using ethylenediaminetetraacetic acid (EDTA), citric acid ((MONO/ANH) and etidronic acid (HEBP) to clean root canals during regenerative endodontic treatments

INTERVENTIONS:
Other: Using ethylenediaminetetraacetic acid (EDTA), citric acid ((MONO/ANH) and etidronic acid (HEBP) to clean root canals during regenerative endodontic treatments — Regenerative endodontic treatment using different irrigation solutions

SUMMARY:
In this study researchers plan to conduct, three different irrigation solutions that are responsible for the release of growth factors necessary for the success of regenerative endodontic treatments will be used. These solutions; Ethylene Diamine Tetra Acetic Acid (EDTA), Etidronic Acid and Citric Acid. The aim of this study is to evaluate the effect of different irrigation solutions used in regenerative endodontic treatment of necrotic open apex molar teeth on postoperative pain. Additionally, the healing of these teeth will be monitored for 1 year.

DETAILED DESCRIPTION:
Root canal treatment is a treatment method applied to milk and permanent teeth. The inflamed and necrotic pulp where the root canal is located is cleaned, debrided chemo-mechanically, and finally filled hermetically with a biocompatible material. Necrotic immature teeth lose their restorative and defensive abilities. Since the root canal walls of these teeth are thin and weak, regenerative endodontic procedures are applied more frequently in the treatment of immature teeth to ensure root development and to restore the vitality of the pulp tissue. In this study researchers plan to conduct, three different irrigation solutions that are responsible for the release of growth factors necessary for the success of regenerative endodontic treatments will be used. These solutions; Ethylene Diamine Tetra Acetic Acid (EDTA), Etidronic Acid and Citric Acid. The aim of this study is to evaluate the effect of different irrigation solutions used in regenerative endodontic treatment of necrotic open apex molar teeth on postoperative pain. Additionally, the healing of these teeth will be monitored for 1 year.

ELIGIBILITY:
Inclusion Criteria:• Molars with open apex

* Teeth with apical periodontitis
* Teeth for which prosthetic restoration is not planned
* Patients between the ages of 8-15 who do not have any significant health problems
* Patients who are not accompanied by periodontal problems and have good oral hygiene

Exclusion Criteria:• People with systemic disease and allergic reactions

* Severely damaged teeth
* If the tooth has previously undergone root canal treatment.
* Use of antibiotics, anti-inflammatory and painkillers in the last two weeks

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 39 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Determining and recording pain levels on the pain scale between treatment sessions | 2 weeks
  Evaluations close to 100 on the postoperative pain scale indicate that the severity of pain increases. Evaluations close to 0 indicate that the severity of pain has decreased.

SECONDARY OUTCOMES:
In the follow-up sessions after the treatment, the size of the lesion in the bone (mm2) is measured by radiography. | 2 years
  Evaluations close to 100 on the scale following lesion healing indicate that the lesion size has increased. Evaluations close to 0 indicate that the lesion size has decreased.

CONTACTS AND LOCATIONS:
Overall Officials: ERASLAN AKYÜZ, Principal Investigator — BAŞ ARAŞTIRMACI; ÜSTÜN, Study Director — YÜRÜTÜCÜ; EMİNSOY AVCI, Study Chair — YARDIMCI ARAŞTIRMACI; SOLAK KOLÇAKOĞLU, Study Chair — YARDIMCI ARAŞTIRMACI; KIZILCI, Study Chair — YARDIMCI ARAŞTIRMACI
Locations (1):
- Erciyes Üniversitesi Diş Hekimliği Fakültesi, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Derived] Akyuz IE, Eminsoy Avci AT, Ustun Y, Kolcakoglu KS, Kizilci E. Evaluation of the effect of different irrigation solutions used in regenerative endodontic treatment of necrotic molar teeth with open apex on postoperative pain- randomized clinical trial. Clin Oral Investig. 2025 Jan 16;29(1):66. doi: 10.1007/s00784-025-06153-3. PMID 39815035